CLINICAL TRIAL: NCT02469051
Title: Usefulness of Breath-hold Triggered SPECT-MPI in Cardiac Hybrid SPECT/CCTA Imaging
Brief Title: Breath-hold Cardiac Hybrid SPECT/CCTA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: USZ-2015-0098
Record Dates: First submitted 2015-05-13; First posted 2015-06-11 (Estimated); Last update posted 2016-05-11 (Estimated); Status verified 2016-05

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Breathhold SPECT-MPI vs. standard freebreathing SPECT-MPI (Other)
  Interventions: Device: Breathhold SPECT-MPI; Device: Standard freebreathing SPECT-MPI; Device: Coronary CT angiography

INTERVENTIONS:
Device: Breathhold SPECT-MPI — Respiratory triggered SPECT myocardial perfusion imaging
Device: Standard freebreathing SPECT-MPI — Clinically indicated, standard non-respiratory triggered SPECT myocardial perfusion imaging
Device: Coronary CT angiography — Clinically indicated coronary CT angiography serving as standard of reference
  Other Names: CCTA

SUMMARY:
This study aims at combining inspiration breath-hold myocardial perfusion SPECT with coronary CT angiography.

ELIGIBILITY:
Inclusion Criteria:

* Referral for cardiac hybrid SPECT/CCTA
* Male and female subjects 18 years of age or older
* Written informed consent by the participant after information about the project

Exclusion Criteria:

* Contraindications for coronary CT angiography (including renal failure with a GFR <30ml/min/1.73m2, allergies to iodinated contrast agents)
* Pregnancy or breast-feeding
* Previous coronary revascularisation
* Inability to follow the examination procedure (e.g. due to language barriers, severe mental disease etc

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2015-05; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Image quality as visually assessed on a Likert scale | 1 day
Number of image artefacts | 1 day

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Nuclear Medicine, University Hospital Zurich, Zurich, Canton of Zurich, Switzerland